CLINICAL TRIAL: NCT04807660
Title: Bacteriological Evaluation of Spontaneous Otorrhea in Children
Brief Title: Bacteriological Evaluation of Children With Otorrhea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Responsible Party: Sponsor
Other Study IDs: ACT0315
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Otorrhea
Keywords: otorrrhea; children; spontaneous perforation of the tympanic membrane; ambulatory; streptococcus pneumoniae; heamophilus influenzae; moraxella catarrhalis; streptococcus pyogenes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective cohort: Middle ear fluid sample for each enrrolled children
  Interventions: Other: middle ear fluid sample

INTERVENTIONS:
Other: middle ear fluid sample — middle ear fluid sample for each enrrolled children

SUMMARY:
After pneumococcal conjugate vaccine implementation, the number of acute otitis media (AOM) episodes has decreased, but AOM still remains among the most common diagnoses in childhood. From 2% to 17% of cases of AOM feature spontaneous perforation of the tympanic membrane (SPTM). The aim of this study was to describe the bacteriological causes of SPTM several years after PCV13 implementation, in 2010.

DETAILED DESCRIPTION:
Since October 2015, children with spontaneous perforation of the tympanic membrane (SPTM) are prospectively enrolled by 41 pediatricians who are part of a research and teaching network (ACTIV, Association Clinique et Thérapeutique Infantile du Val de Marne [Clinical and Therapeutic Association of Val de Marne]) throughout France. For some patients, otorrhea is the first manifestation of AOM; for others, otorrhea occurred after AOM treatment failure or recurrence. Failure (non-responsive AOM) is defined as otorrhea appearing despite at least 48 hr of antibiotics or recurring less than 4 days after the end of antibiotic treatment. Recurrence is defined by the appearance of otorrhea 4 to 30 days after the end of antibiotic treatment for AOM.

Middle ear fluid (MEF) is obtained by sampling spontaneous discharge according to clinical practice guidelines. MEF specimens are obtained with cotton-tipped wire swabs, immediately placed in transport medium (Copan Venturi Transystem®, Brescia, Italy), and transported within 48 hr to one of the two centralized microbiology laboratories (Robert Debré Hospital or National Centre for Pneumococci at European Georges Pompidou Hospital, Paris, France).

ELIGIBILITY:
Inclusion Criteria:

* children from 3 months to 15 years old
* with otorrhea
* signed parents consent

Exclusion Criteria:

* children under 3 months
* children > 15 years old

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all children from 3 months to 15 years old with otorrhea
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Bacteria identification | at inclusion
  The percentage of children with otopathogens

SECONDARY OUTCOMES:
Describe the serotypes of S. pneumoniae | at inclusion
  percentage of each serotype
Describe the resistance of heamophilus influenzae | at inclusion
  percentage of resistant h. inlfuenzae

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cohen, Study Director — Association Clinique et Thérapeutique Infantile du Val de Marne
Locations (1):
- ACTIV, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cohen R, Varon E, Bidet P, Cohen JF, Bechet S, Couloigner V, Michot AS, Guiheneuf C, Bonacorsi S, Levy C. Diagnostic Accuracy of Group A Streptococcus Rapid Antigen Detection Test on Middle Ear Fluid in Children With Acute Otitis Media With Spontaneous Perforation: A Prospective Multicenter Evaluation. Pediatr Infect Dis J. 2023 Sep 1;42(9):816-818. doi: 10.1097/INF.0000000000004009. Epub 2023 Jun 22. PMID 37368992
- See also: Bacterial causes of otitis media with spontaneous perforation of the tympanic membrane in the era of 13 valent pneumococcal conjugate vaccine — https://pubmed.ncbi.nlm.nih.gov/30707730/